CLINICAL TRIAL: NCT01730053
Title: A Randomized, Double-Blind Study of the Efficacy and Safety of REGN727 Added-on to Rosuvastatin Versus Ezetimibe Added-on to Rosuvastatin Versus Rosuvastatin Dose Increase in Patients Who Are Not Controlled on Rosuvastatin
Brief Title: Study of Alirocumab (REGN727/SAR236553) added-on to Rosuvastatin Versus Other Lipid Modifying Treatments (LMT) (ODYSSEY OPTIONS II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R727-CL-1118
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Rosuvastatin 20 mg (Active Comparator): Participants, who were receiving rosuvastatin 10 mg over-encapsulated tablet orally at baseline, received rosuvastatin 20 mg over-encapsulated tablet orally once daily (QD), placebo for alirocumab SC injection every two weeks (Q2W), and placebo for ezetimibe over-encapsulated tablet orally QD added to stable Lipid-Modifying Therapy (LMT) for 24 weeks.
  Interventions: Drug: Rosuvastatin; Drug: Placebo
- Ezetimibe 10 mg + Rosuvastatin 10 mg (Active Comparator): Participants, who were receiving rosuvastatin 10 mg over-encapsulated tablet orally at baseline, received ezetimibe 10 mg over-encapsulated tablet orally QD, rosuvastatin 10 mg over-encapsulated tablet orally QD, and placebo for alirocumab SC injection Q2W added to stable LMT for 24 weeks.
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe; Drug: Placebo
- Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg (Experimental): Participants, who were receiving rosuvastatin 10 mg over-encapsulated tablet orally at baseline, received alirocumab 75 mg SC injection Q2W, rosuvastatin 10 mg over-encapsulated tablet orally QD, and placebo for ezetimibe over-encapsulated tablet orally QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
  Interventions: Drug: Alirocumab; Drug: Rosuvastatin; Drug: Placebo
- Rosuvastatin 40 mg (Active Comparator): Participants, who were receiving rosuvastatin 20 mg over-encapsulated tablet orally at baseline, received rosuvastatin 40 mg over-encapsulated tablet orally QD, placebo for alirocumab Q2W SC injection, and placebo for ezetimibe QD over-encapsulated tablet orally added to stable LMT for 24 weeks.
  Interventions: Drug: Rosuvastatin; Drug: Placebo
- Ezetimibe 10 mg + Rosuvastatin 20 mg (Active Comparator): Participants, who were receiving rosuvastatin 20 mg over-encapsulated tablet orally at baseline, received ezetimibe 10 mg over-encapsulated tablet orally QD, rosuvastatin 20 mg over-encapsulated tablet orally QD, and placebo for alirocumab Q2W SC injection added to stable LMT for 24 weeks.
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe; Drug: Placebo
- Alirocumab 75 mg/ up to 150 mg + Rosuvastatin 20 mg (Experimental): Participants, who were receiving rosuvastatin 20 mg over-encapsulated tablet orally at baseline, received alirocumab 75 mg Q2W SC injection, rosuvastatin 20 mg over-encapsulated tablet orally QD, and placebo for ezetimibe over-encapsulated tablet orally QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
  Interventions: Drug: Alirocumab; Drug: Rosuvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Alirocumab — Alirocumab administered as a SC injection of 1 mL into the abdomen, thigh, or outer area of the upper arm.
  Other Names: REGN727/SAR236553
  Arms: Alirocumab 75 mg/ up to 150 mg + Rosuvastatin 20 mg; Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg
Drug: Rosuvastatin — Rosuvastatin over-encapsulated tablets orally.
  Other Names: Crestor
Drug: Ezetimibe — Ezetimibe over-encapsulated tablets orally.
  Other Names: Ezetrol
  Arms: Ezetimibe 10 mg + Rosuvastatin 10 mg; Ezetimibe 10 mg + Rosuvastatin 20 mg
Drug: Placebo — Placebo for alirocumab and ezetimibe.

SUMMARY:
To evaluate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab (REGN727/SAR236553) as an add-on therapy to other LMT in patients with hypercholesterolemia at high cardiovascular (CV) risk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with LDL-C greater than or equal to 70 mg/dL at the screening visit and who are not adequately controlled with a stable daily dose of rosuvastatin, with or without other LMT.

   OR
2. Patients with screening LDL-C greater than or equal to 100 mg/dL who are not adequately controlled with a stable daily dose of rosuvastatin before the screening visit, with or without other LMT.

Exclusion Criteria:

1. LDL-C less than 70 mg/dL at the screening visit in patients with history of documented cardiovascular disease (CVD)
2. LDL-C less than 100 mg/dL at the screening visit in patients without history of documented coronary heart disease (CHD) or non-CHD CVD, but with other risk factors
3. Homozygous familial hypercholesterolemia (FH) (clinically or previous genotyping)
4. Recent (within 3 months prior to the screening visit) myocardial infarction (MI), unstable angina leading to hospitalization, percutaneous coronary intervention (PCI), coronary bypass graft surgery (CABG), uncontrolled cardiac arrhythmia, stroke, transient ischemic attack, carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease
5. Newly diagnosed (within 3 months prior to randomization visit) or poorly controlled diabetes
6. Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins

(The inclusion/ exclusion criteria provided above is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (93):
- United States (54):
  - Chandler, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Beverly Hills, California
  - Fair Oaks, California
  - Newport Beach, California
  - Northridge, California
  - Sacramento, California
  - Walnut Creek, California
  - Milford, Connecticut
  - Atlantis, Florida
  - Bradenton, Florida
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Lakeland, Florida
  - (2 Locations), Miami, Florida
  - Oviedo, Florida
  - Pinellas Park, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Boise, Idaho
  - Morton, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newton, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Auburn, Maine
  - Bethesda, Maryland
  - Edina, Minnesota
  - Rochester, Minnesota
  - Olive Branch, Mississippi
  - Port Gibson, Mississippi
  - St Louis, Missouri
  - Butte, Montana
  - Williamsville, New York
  - Cincinnati, Ohio
  - Marion, Ohio
  - Portland, Oregon
  - Warwick, Rhode Island
  - Greer, South Carolina
  - Summerville, South Carolina
  - Kingsport, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Bountiful, Utah
  - Salt Lake City, Utah
- Australia (5):
  - Herston
  - New Lambton Heights
  - Perth
  - Sherwood
  - Woolloongabba
- Canada (8):
  - Brampton, Ontario
  - Burlington, Ontario
  - Etobicoke, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
- France (2):
  - Dijon
  - Lille
- Germany (5):
  - Bad Oeynhausen
  - Berlin
  - Cologne
  - Regensburg
  - Ulm
- Italy (5):
  - Chieti
  - Genova
  - Napoli
  - Palermo
  - (2 Locations), Roma
- Mexico (5):
  - Baja California
  - Distrito Federal
  - (3 Locations), Guadalajara
  - Monterrey
  - Zapopan Jalisco
- Spain (4):
  - (2 Locations), Barcelona
  - Madrid
  - Santiago
  - Seville
- United Kingdom (5):
  - West Bromwich, West Midlands
  - Chester
  - Peterborough
  - Salford
  - Stevenage

REFERENCES:
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279
- [Derived] Farnier M, Jones P, Severance R, Averna M, Steinhagen-Thiessen E, Colhoun HM, Du Y, Hanotin C, Donahue S. Efficacy and safety of adding alirocumab to rosuvastatin versus adding ezetimibe or doubling the rosuvastatin dose in high cardiovascular-risk patients: The ODYSSEY OPTIONS II randomized trial. Atherosclerosis. 2016 Jan;244:138-46. doi: 10.1016/j.atherosclerosis.2015.11.010. Epub 2015 Nov 14. PMID 26638010
- [Derived] Robinson JG, Colhoun HM, Bays HE, Jones PH, Du Y, Hanotin C, Donahue S. Efficacy and safety of alirocumab as add-on therapy in high-cardiovascular-risk patients with hypercholesterolemia not adequately controlled with atorvastatin (20 or 40 mg) or rosuvastatin (10 or 20 mg): design and rationale of the ODYSSEY OPTIONS Studies. Clin Cardiol. 2014 Oct;37(10):597-604. doi: 10.1002/clc.22327. Epub 2014 Sep 30. PMID 25269777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 79 sites in 8 countries. Overall, 672 participants were screened between 24 October 2012 and 27 September 2013, 367 of whom were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction or ischemic stroke, and intensity of statin treatment (rosuvastatin 10 or 20 mg). Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System (IVWRS) in a 1:1:1:1:1:1 ratio after confirmation of selection criteria.
Groups:
- Rosuvastatin 20 mg: Participants who were receiving rosuvastatin 10 mg at baseline, received rosuvastatin 20 mg once daily (QD), placebo for alirocumab every 2 weeks (Q2W), and placebo for ezetimibe QD added to stable lipid-modifying therapy (LMT) for 24 weeks.
- Ezetimibe 10 mg + Rosuvastatin 10 mg: Participants who were receiving rosuvastatin 10 mg at baseline, received ezetimibe 10 mg QD, rosuvastatin 10 mg QD, and placebo for alirocumab Q2W added to stable LMT for 24 weeks.
- Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg: Participants who were receiving rosuvastatin 10 mg at baseline, received alirocumab 75 mg Q2W, rosuvastatin 10 mg QD, and placebo for ezetimibe QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when low-density lipoprotein cholesterol (LDL-C) levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
- Rosuvastatin 40 mg: Participants who were receiving rosuvastatin 20 mg at baseline, received rosuvastatin 40 mg QD, placebo for alirocumab Q2W, and placebo for ezetimibe QD added to stable LMT for 24 weeks.
- Ezetimibe 10 mg + Rosuvastatin 20 mg: Participants who were receiving rosuvastatin 20 mg at baseline, received ezetimibe 10 mg QD, rosuvastatin 20 mg QD, and placebo for alirocumab Q2W added to stable LMT for 24 weeks.
- Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg: Participants who were receiving rosuvastatin 20 mg at baseline, received alirocumab 75 mg Q2W, rosuvastatin 20 mg QD, and placebo for ezetimibe QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
Period: Overall Study
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Started | 48 | 48 | 49 | 53 | 53 | 54
Treated | 48 | 48 | 49 | 53 | 53 | 54
Completed | 43 | 34 | 38 | 45 | 44 | 41
Not Completed | 5 | 14 | 11 | 8 | 9 | 13
Not completed — Participant moved | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 6 | 3 | 3 | 2 | 2
Not completed — Poor compliance to protocol | 1 | 2 | 2 | 0 | 0 | 2
Not completed — Other than specified | 2 | 6 | 5 | 4 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Alirocumab 75/up to 150 + Rosuvastatin 10 mg: Participants, who were receiving rosuvastatin 10 mg over-encapsulated tablet orally at baseline, received alirocumab 75 mg SC injection Q2W, rosuvastatin 10 mg over-encapsulated tablet orally QD, and placebo for ezetimibe over-encapsulated tablet orally QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75/up to 150 + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg | Total
Number analyzed (Participants) | 48 | 48 | 49 | 53 | 53 | 54 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.15) | 60.4 (10.38) | 62.2 (11.11) | 60.6 (10.11) | 63.1 (10.2) | 57.9 (8.86) | 60.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 18 | 15 | 22 | 26 | 118
  Male | 33 | 26 | 31 | 38 | 31 | 28 | 187
Low density lipoprotein cholesterol (LDL-C) in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C from Friedewald formula.
  mg/dL | 105.9 (36.0) | 102.4 (41.9) | 107.3 (26.4) | 112.9 (43.3) | 119.0 (48.0) | 118.3 (32.2) | 111.3 (39.0)
LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C from Friedewald formula.
  mmol/L | 2.743 (0.933) | 2.653 (1.085) | 2.78 (0.684) | 2.924 (1.122) | 3.082 (1.243) | 3.065 (0.834) | 2.882 (1.009)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT) Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -16.3 (4.1) | -14.4 (4.4) | -50.6 (4.2) | -15.9 (7.1) | -11.0 (7.2) | -36.3 (7.1)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Alirocumab group was compared to the corresponding active control group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -34.2, 98.75% CI 2-sided [-49.2 to -19.3]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; As described in statistical analysis 1 of the endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -36.1, 98.75% CI 2-sided [-51.5 to -20.7]
Statistical Analysis 3: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg; As described in statistical analysis 1 of the endpoint; Test type: Superiority or Other; p = 0.0453, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -20.3, 98.75% CI 2-sided [-45.8 to 5.1]
Statistical Analysis 4: Comparison: Ezetimibe 10 mg + Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg; As described in statistical analysis 1 of the endpoint; Test type: Superiority or Other; p = 0.0136, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -25.3, 98.75% CI 2-sided [-50.9 to 0.3]

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (ie. up to 21 days after last injection or 3 days after the last capsule [whatever rosuvastatin or ezetimibe], whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 46 | 48 | 50 | 50 | 51
percent change | -18.3 (3.3) | -20.3 (3.6) | -53.5 (3.5) | -17.0 (6.9) | -16.5 (6.9) | -41.5 (6.9)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 1.25 % level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -35.2, 98.75% CI 2-sided [-47.4 to -23.0]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -33.2, 98.75% CI 2-sided [-45.9 to -20.5]
Statistical Analysis 3: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0131, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -24.5, 98.75% CI 2-sided [-49.2 to 0.2]

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment (ITT analysis).
Time Frame: From Baseline to Week 12
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -17.1 (4.1) | -17.4 (4.2) | -49.6 (4.1) | -22.1 (5.3) | -19.3 (5.4) | -32.3 (5.2)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant for rosuvastatin 10 mg baseline stratification); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -35.2, 98.75% CI 2-sided [-47.4 to -17.9]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -32.2, 98.75% CI 2-sided [-47 to -17.5]

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule [whatever rosuvastatin or ezetimibe], whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 12
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 46 | 48 | 50 | 50 | 51
percent change | -17.2 (3.6) | -20.3 (3.8) | -52.6 (3.6) | -22.9 (5.2) | -21.8 (5.2) | -35.1 (5.2)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -35.3, 98.75% CI 2-sided [-48.2 to -22.5]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -32.3, 98.75% CI 2-sided [-45.6 to -19.0]

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 44 | 44 | 44 | 51 | 48 | 49
percent change | -7.3 (3.0) | -9.7 (3.1) | -36.5 (3.1) | -9.8 (4.1) | -11.2 (4.3) | -28.3 (4.3)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -29.2, 98.75% CI 2-sided [-40.1 to -18.3]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -26.8, 98.75% CI 2-sided [-37.9 to -15.7]

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (ie. up to 21 days after last injection or 3 days after the last capsule [whatever rosuvastatin or ezetimibe], whichever came first).
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 44 | 42 | 43 | 50 | 47 | 48
percent change | -8.8 (2.6) | -11.2 (2.7) | -39.5 (2.6) | -12.7 (4.0) | -12.6 (4.1) | -30.4 (4.2)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -30.7, 98.75% CI 2-sided [-40.1 to -21.3]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -28.3, 98.75% CI 2-sided [-38.0 to -18.7]

7. Secondary Outcome: Percent Change From Baseline in Non-High-density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -11.3 (3.4) | -13.4 (3.7) | -42.7 (3.5) | -11.2 (5.1) | -12.9 (5.2) | -31.4 (5.2)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -31.4, 98.75% CI 2-sided [-43.9 to -18.9]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -29.3, 98.75% CI 2-sided [-42.1 to -16.4]

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule [whatever rosuvastatin or ezetimibe], whichever came first).
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the mITT population with one baseline and at least one post-baseline Non-HDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 46 | 48 | 50 | 50 | 51
percent change | -12.9 (2.8) | -17.5 (3.1) | -45.7 (2.9) | -14.9 (4.2) | -18.2 (4.2) | -35.6 (4.3)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -32.8, 98.75% CI 2-sided [-43.2 to -22.4]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -28.2, 98.75% CI 2-sided [-39.1 to -17.3]

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -8.3 (2.4) | -8.7 (2.6) | -28.9 (2.5) | -8.5 (3.6) | -12.4 (3.6) | -20.6 (3.6)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -20.6, 98.75% CI 2-sided [-29.4 to -11.8]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -20.3, 98.75% CI 2-sided [-29.3 to -11.2]

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 44 | 44 | 44 | 51 | 48 | 49
percent change | -8.1 (3.2) | -12.1 (3.3) | -36.1 (3.2) | -13.7 (3.3) | -14.3 (3.3) | -29.0 (3.3)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -28.1, 98.75% CI 2-sided [-39.7 to -16.5]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -24.0, 98.75% CI 2-sided [-35.7 to -12.3]

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 12
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -11.7 (3.5) | -16.3 (3.6) | -41.2 (3.5) | -18.0 (3.6) | -18.7 (3.7) | -29.8 (3.6)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -29.5, 98.75% CI 2-sided [-42.1 to -16.9]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -24.9, 98.75% CI 2-sided [-37.7 to -12.2]

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 12
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/ up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -8.9 (2.6) | -11.8 (2.7) | -29.0 (2.6) | -13.8 (2.8) | -13.9 (2.8) | -19.4 (2.7)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -20.1, 98.75% CI 2-sided [-29.4 to -10.7]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.0125; LS Mean Difference = -17.2, 98.75% CI 2-sided [-26.7 to -7.7]

13. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - ITT Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted percentages at Week 24 were obtained from a multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to week 24 regardless of status on- or off-treatment were included in the imputation model (ITT analysis).
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percentage of participants | 45.0 | 57.2 | 84.9 | 40.1 | 52.2 | 66.7
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant for rosuvastatin 10 mg baseline stratification). Statistical analysis used a multiple imputation approach followed by a Logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 12.4, 98.75% CI 2-sided [2.6 to 59.5]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0007, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 8.4, 98.75% CI 2-sided [1.8 to 40.5]

14. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted percentages at Week 24 were obtained from a multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 24 i.e. up to 21 days after last injection or 3 days after the last capsule [whatever rosuvastatin or ezetimibe], whichever came first (on-treatment analysis).
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 46 | 48 | 50 | 50 | 51
percentage of participants | 47.0 | 60.5 | 86.4 | 41.3 | 54.8 | 70.4
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 15.6, 98.75% CI 2-sided [2.58 to 88.2]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 9.9, 98.75% CI 2-sided [1.7 to 56.7]

15. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: as for outcome 13
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percentage of participants | 31.3 | 43.1 | 77.8 | 29.9 | 43.6 | 60.1
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 18.6, 98.75% CI 2-sided [3.6 to 96.2]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 11.6, 98.75% CI 2-sided [2.5 to 53.1]

16. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: as for outcome 14
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 46 | 48 | 50 | 50 | 51
percentage of participants | 34.8 | 46.7 | 76.5 | 30.6 | 45.1 | 66.1
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 20.3, 98.75% CI 2-sided [2.4 to 67.7]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0002, Regression, Logistic — Threshold for significance ≤ 0.0125; Odds Ratio (OR) = 12.7, 98.75% CI 2-sided [2.4 to 67.7]

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from a multiple imputation approach model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/ up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -4.0 (4.3) | -4.3 (4.5) | -27.9 (4.1) | -5.2 (4.8) | -5.8 (4.6) | -22.7 (5.1)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant for rosuvastatin 10 mg baseline stratification). Statistical analysis used a multiple imputation approach followed by a robust regression model; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.0125; Adjusted Mean Difference = -23.9, 98.75% CI 2-sided [-38.6 to -9.1]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Rosuvastatin 10 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0001, Regression, Robust — Threshold for significance ≤ 0.0125; Adjusted Mean Difference = -23.6, 98.75% CI 2-sided [-39.0 to -8.2]

18. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | 1.7 (2.4) | 4.0 (2.5) | 9.1 (2.4) | 1.5 (2.3) | -1.8 (2.3) | 7.2 (2.3)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.0311, Regression, Robust — Threshold for significance ≤ 0.0125; LS Mean Difference = 7.4, 98.75% CI 2-sided [-1.2 to 16.1]

19. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: as for outcome 17
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -1.8 (4.5) | -8.3 (4.8) | -11.2 (4.6) | -9.9 (4.1) | -11.1 (4.3) | -8.7 (4.5)

20. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 44 | 44 | 44 | 51 | 48 | 49
percent change | 5.4 (1.9) | 5.0 (1.9) | 6.7 (1.9) | 2.9 (1.9) | -0.9 (1.9) | 6.7 (2.0)

21. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from a multiple imputation approach model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 12
Population: Lipoprotein (a) ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | -0.7 (3.5) | -3.9 (3.6) | -20.7 (3.5) | 3.5 (4.2) | 7.9 (4.1) | -16.0 (4.2)

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 12
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | 0.7 (2.1) | 0.2 (2.2) | 5.9 (2.1) | 0.6 (2.5) | 3.1 (2.5) | 8.0 (2.5)

23. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 21
Time Frame: From Baseline to Week 12
Population: Fasting triglycerides ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 48 | 47 | 48 | 52 | 50 | 53
percent change | 8.1 (4.1) | -8.2 (4.2) | -14 (4.1) | -2.7 (4.0) | -12.4 (4.0) | -10.1 (4.0)

24. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 12
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Number analyzed (Participants) | 44 | 44 | 44 | 51 | 48 | 49
percent change | 4.0 (1.6) | 2.6 (1.6) | 4.3 (1.6) | 0.9 (1.8) | 1.8 (1.8) | 9.1 (1.8)

ADVERSE EVENTS:
Time Frame: From Baseline to Week 32
Description: Treatment emergent adverse events that developed during on-treatment period (the time period from the first double-blind injection of study drug up to the day of last injection + 70 days) are reported.
Arm/Group | Rosuvastatin 20 mg | Ezetimibe 10 mg + Rosuvastatin 10 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Rosuvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg
Serious Adverse Events (participants affected / at risk) | 4/48 | 5/48 | 2/49 | 4/53 | 3/53 | 4/54
Other Adverse Events (participants affected / at risk) | 11/48 | 11/48 | 11/49 | 20/53 | 12/53 | 15/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin 20 mg (N=48) | Ezetimibe 10 mg + Rosuvastatin 10 mg (N=48) | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg (N=49) | Rosuvastatin 40 mg (N=53) | Ezetimibe 10 mg + Rosuvastatin 20 mg (N=53) | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg (N=54)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin 20 mg (N=48) | Ezetimibe 10 mg + Rosuvastatin 10 mg (N=48) | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 10 mg (N=49) | Rosuvastatin 40 mg (N=53) | Ezetimibe 10 mg + Rosuvastatin 20 mg (N=53) | Alirocumab 75 mg/up to 150 mg + Rosuvastatin 20 mg (N=54)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 6 (6) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 6 (7) | 4 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 5 (5) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.